CLINICAL TRIAL: NCT05609916
Title: CBT Augmentation to Promote Medication Discontinuation in Pediatric OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-52089
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Behavioral Therapy; Obsessive-Compulsive Disorder; Obsessive-Compulsive Disorder in Children; Obsessive-Compulsive Disorder in Adolescence
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continued SRI (Active Comparator): After post-phase I assessment, participants who are eligible will be randomized to 1) Continued SRI. For these participants, the medication (SRI) will be provided at a consistent dosage.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Discontinuation titration to placebo (Placebo Comparator): After post-phase I assessment, participants who are eligible will be randomized to 2) Discontinuation titration to placebo. For these participants, the placebo substitution in an increasing proportion of capsules will be implemented until all drug is withdrawn.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Open label CBT (Other): During Phase I, all participants will receive open label cognitive-behavioral therapy. Only those who achieve significant benefit will be able to most on to the post-phase I assessment, and then to the random assignment to Continued SRI or Discontinuation titration to placebo arms.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — During Phase I, participants will receive open label (no blinding) CBT during their study participation for 12 to 18 weeks.
  During Phase II, participants will continue receiving CBT maintenance sessions every two weeks for the first 4 weeks, followed by sessions every four weeks. They will also meet with the study physician every 2 weeks via telepsychiatry appointments for clinical and scalar assessment.

SUMMARY:
The purpose of this study is to examine whether youth with OCD who benefit from CBT augmentation to SRI can discontinue their medication without relapse over 24 weeks.

DETAILED DESCRIPTION:
Pediatric obsessive-compulsive disorder (OCD) is a common, chronic, and severe psychiatric disorder. Currently, many youth with OCD are treated with medication, such as a serotonin reuptake inhibitor (SRI); however, only a subset of them responds to SRI. Data show that the addition of cognitive-behavioral therapy (CBT) to SRI partial responders is effective although extended SRI use with CBT can attenuate combined treatment outcomes. This placebo-controlled study will enroll pediatric OCD patients to examine if those who benefit from CBT augmentation can discontinue their SRI successfully without relapse over 24-weeks. This study will also bank genomic samples for future analysis when polygenic risk scores for OCD may become available.

This study will be conducted in two phases. In Phase I, all participants will receive a web-based CBT for 12 to 18 weeks. At the end of Phase I, those who achieve wellness indicated by CY-BOCS ≤ 12 and ≥ 50% reduction since baseline for 3 consecutive weeks, will go on to the next phase. In Phase II, participants will be randomized into two groups: 1) Continued SRI and 2) Discontinuation titration to placebo. In this phase, all participants will receive web-based CBT maintenance sessions and attend medication visits for 24 weeks. At 12 months after the end of Phase II, all participants will complete a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7 to 17 at enrollment with a primary diagnosis of OCD of > 6 months duration based on the Kiddie Schedule for Affective Disorders and Schizophrenia Lifetime Version for DSM-5 (KSADS-PL) and have a CY-BOCS ≥ 16.
* The child is on stable and maximally tolerated SRI medication (i.e., clomipramine, fluoxetine, fluvoxamine, sertraline, citalopram, escitalopram) for ≥12 weeks given that they are persistently and moderately symptomatic. Paroxetine is exclusionary due to safety concerns.
* Both the child and parent participating in the study are English speaking.
* Both the child and their parent participating in the study reside in Texas.

Exclusion Criteria:

* The child has a diagnosis of lifetime DSM-5 bipolar disorder, psychotic disorder, and/or intellectual disability.
* The child has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention.
* The child is receiving concurrent psychotherapy for OCD.
* Initiation of a psychotropic medication less than 4 weeks prior to study enrollment or a stimulant/psychoactive medication less than 2 weeks prior to study enrollment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | 7 days
  Clinician-rated child OCD symptoms and severity throughout the past week. The scale has a checklist of obsessions and compulsions, followed by severity items each scored on a 0 to 4 scale.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement | 7 days
  Clinician-rated child psychopathology improvement since initial rating. A single item is scored 0-6 (0 = very much worse; 6 = very much improved).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No